CLINICAL TRIAL: NCT03693859
Title: Smart Gaming for Obesity: A Randomized Trial
Brief Title: Smart Gaming in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lent1018
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Weight Loss + Gaming (Experimental): Treatment will consist of 12-weekly, one-hour group sessions of approximately 15 participants per group. Participants will provide logs of serious gaming (intervention).
  Interventions: Behavioral: Cognitive enhancement program
- Behavioral Weight Loss + Health Segments (Active Comparator): Control participants will be asked to spend 30 minutes watching health segments online, five days per week, for 8 weeks. Participants will provide logs of video segment watching (control).
  Interventions: Behavioral: Behavioral Weight Loss + Health Segments

INTERVENTIONS:
Behavioral: Cognitive enhancement program — The cognitive enhancement condition (BWL+GAMING) will both teach the behavioral skills necessary for weight loss and strengthen the executive functions that underlie these skills.
  Other Names: Smart Gaming
  Arms: Behavioral Weight Loss + Gaming
Behavioral: Behavioral Weight Loss + Health Segments — Control participants will be asked to spend 30 minutes watching health segments online, five days per week, for 8 weeks.
  Arms: Behavioral Weight Loss + Health Segments

SUMMARY:
Obesity (Body Mass Index ≥ 30 kg/m2) is associated with diminished executive functioning. The primary objective of this randomized, controlled trial is to evaluate the efficacy of a behavioral weight loss program coupled with enhanced executive functioning training via serious gaming on weight loss and weight loss maintenance in adults with obesity and executive functioning deficits compared to adults undergoing standard behavioral treatment alone (N = 200). Serious gaming interventions that target the specific cognitive functions needed for weight-loss maintenance may improve long-term weight-loss success.

DETAILED DESCRIPTION:
This randomized, controlled study will evaluate the efficacy of a behavioral weight loss program coupled with enhanced executive functioning training via serious gaming (BWL+GAMING) on weight loss and maintenance in adults with obesity and executive functioning deficits compared to standard behavioral treatment alone (BWL) at two urban Philadelphia university-based clinics (PCOM [Philadelphia College of Osteopathic Medicine] and Temple University). Participants will be recruited from the community. All participants (N = 200) will complete 12 weeks of behavioral weight loss treatment. Intervention participants will also complete 30-minutes (5 days per week for 8 weeks) of a serious gaming program, which will feature online games developed specifically to enhance executive functions. The primary outcomes are weight change and weight change maintenance, which will be measured at 12 and 52 weeks, respectively. Neuropsychological testing will evaluate the proposed mechanism of action, changes in executive functioning, before and after treatment (12 and 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Executive functioning deficits
* Internet access

Exclusion Criteria:

* Under 18 years of age
* Over 65 years of age
* Taking weight loss medication
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Weight change | 52 weeks
  Weight change maintenance of at least 5%

IPD SHARING:
Plan to Share IPD: Undecided